CLINICAL TRIAL: NCT02583711
Title: The Step Home Trial: Utilising Physical Activity Data in the Acute Post-operative Setting
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 15SM2689; 15/LO/1038 (Other: NRES London City Road & Hampstead)
Record Dates: First submitted 2015-09-30; First posted 2015-10-22 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Surgery; Enhanced Recovery; Technology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Activity sensor (3 axis accelerometer) — Patient cohort will wear the activity sensor from pre-admission clinic until discharge after surgical procedure

SUMMARY:
This is an observational study, which aims to assess how physical activity levels following surgical procedures correlate with patient recovery and length of hospital stay, as well as the utility of this physical activity data to the postoperative surgical team. Surgical teams frequently enquire about their patients' physical activity levels on postoperative ward rounds. Although this information is often provided anecdotally by nursing staff and junior doctors, there are no objective data made available to the clinician. Such data has the potential to supplement other observations (e.g. heart rate, blood pressure, temperature) to help gain an impression of a patient's recovery and physical status, this in turn could provide evidence to help facilitate early discharge as well as to predict medium to longterm outcomes. Advances in wearable technology allow the investigators to collect detailed information with regard to activity with minimal disruption.

Recent literature has shown that these wristworn sensors can feasibly be worn in hospital pre and postoperatively, with evidence of a correlation between the amount of steps taken postoperatively and the length of hospital stay. This study will provide further evidence for the usability and utility of wearable sensors in the inpatient surgical setting. It will provide supporting evidence for surgeons to confidently analyse and assess patients in hospital, allowing for safe and expedient discharge home as well as identify highrisk patients who are likely to require extra support and surveillance in the community setting.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective surgical operative procedure

Exclusion Criteria:

* Unable to mobilise independently Have medical condition characterized by movement disorder e.g. Parkinson's Disease Unable to understand and complete the SF-36 (unless interpreter present) or lack capacity to consent Psychological Disorder Aged less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients due for elective surgical procedures will be recruited from outpatient general surgical clinic
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Hospital, London, Not in US/Canada, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Cohort: Normal healthy cohort not undergoing colorectal surgical management
- Patients Wearing WAM Pre-op and Post-op on the Ward: Patients who underwent colorectal surgery and wore a wearable activity monitor at home pre-operatively and also post-operatively on the ward until discharge
- Patients Who Wore WAM Pre-op, Post-op on the Ward and Home: Patients who underwent colorectal surgery and wore a wearable activity monitor both pre-operatively, and post-operatively both on the ward and at home.
Period: Overall Study
Arm/Group | Healthy Cohort | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Started | 11 | 38 | 10
Completed | 11 | 28 | 10
Not Completed | 0 | 10 | 0
Not completed — Withdrawal by Subject | 0 | 10 | 0

BASELINE CHARACTERISTICS:
Population: Only 28 patients in the Pre-op/post-op group completed the study, 10 participants did not have full data available for analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Cohort | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home | Total
Number analyzed (Participants) | 11 | 28 | 10 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.26) | 67 (11.2) | 65 (9.2) | 66 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 16 | 5 | 27
  Male | 5 | 12 | 5 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 28 | 10 | 49

OUTCOME MEASURES:

1. Primary Outcome: Total Activity Pre-op
Time Frame: 2-3 weeks
Measure: Mean (Standard Deviation); unit: minutes of activity per 24 hour period
Arm/Group | Healthy Cohort | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Number analyzed (Participants) | 11 | 28 | 10
minutes of activity per 24 hour period | 177 (43) | 154 (88) | 186 (73)

2. Primary Outcome: Length of Hospital Stay
Time Frame: hospital stay (through hospital stay, approximately to 35 days)
Measure: Median (Full Range); unit: days
Arm/Group | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Number analyzed (Participants) | 28 | 10
days | 7 [3 to 33] | 8 [4 to 13]

3. Primary Outcome: Time Spent in Light Activity - Pre-op
Description: Signal vector magnitude (SVM) and cut point analysis algorithms are used with the tri-axial accelerometer data to quantify activity into sedentary, light, moderate and vigorous activity.
  The time spent in the different activity levels was analysed from the recorded accelerometer data and analysed.
Time Frame: 2-3 weeks
Measure: Mean (Standard Deviation); unit: minutes of activity per 24 hour period
Arm/Group | Healthy Cohort | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Number analyzed (Participants) | 11 | 28 | 10
minutes of activity per 24 hour period | 95 (24) | 75 (41) | 87 (38)

4. Primary Outcome: Time Spent in Moderate Activity - Preop
Description: as for outcome 3
Time Frame: 2-3 weeks
Measure: Mean (Standard Deviation); unit: minutes of activity per 24 hour period
Arm/Group | Healthy Cohort | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Number analyzed (Participants) | 11 | 28 | 10
minutes of activity per 24 hour period | 87 (25) | 80 (56) | 98 (40)

5. Primary Outcome: Time Spent in Vigorous Activity - Pre-op
Description: as for outcome 3
Time Frame: 2-3 weeks
Measure: Mean (Standard Deviation); unit: minutes of activity per 24 hour period
Arm/Group | Healthy Cohort | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Number analyzed (Participants) | 11 | 28 | 10
minutes of activity per 24 hour period | 0 (0) | 0 (1) | 0 (1)

6. Secondary Outcome: Number of Participants With Re-admission at Day 30
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Number analyzed (Participants) | 28 | 10
Participants | 3 | 1

7. Secondary Outcome: Number of Participants With Complications up to 6 Weeks Post Discharge
Time Frame: up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
Number analyzed (Participants) | 28 | 10
Participants | 10 | 4

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Healthy Cohort | Patients Wearing WAM Pre-op and Post-op on the Ward | Patients Who Wore WAM Pre-op, Post-op on the Ward and Home
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/28 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/28 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/28 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02583711/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02583711/ICF_001.pdf